CLINICAL TRIAL: NCT02902978
Title: A Phase 1 Single Dose Study of E6130 in Japanese Healthy Adult Male Subjects
Brief Title: A Single Dose Study of E6130 in Japanese Healthy Adult Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EA Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: E6130-J081-001
Record Dates: First submitted 2016-09-13; First posted 2016-09-16 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2017-09

CONDITIONS: Japanese Healthy Adult Male Participants
Keywords: E6130; Japanese healthy adult male participants; Phase 1; Pharmacokinetics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 to 7 (Experimental): Participants will receive a single dose of E6130 or placebo, administered in a dose-ascending manner under the fasted condition.
  Interventions: Drug: E6130; Drug: Placebo
- Cohort 8 (Experimental): Participants will receive a single dose of E6130 (determined in Cohort 1 to 7), administered in the specified order (fed/fasted or fasted/fed) to evaluate the food effect.
  Interventions: Drug: E6130

INTERVENTIONS:
Drug: E6130
Drug: Placebo — E6130 matched placebo
  Arms: Cohort 1 to 7

SUMMARY:
The primary purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics of a single dose of E6130 in Japanese healthy adult male participants.

DETAILED DESCRIPTION:
This study consists of 8 cohorts, Cohorts 1 to 8. Cohorts 1 to 7 are designed as a single-center, single dose, placebo-controlled, randomized, ascending dose, double-blind study. Cohort 8 is designed as a single-center, single dose, randomized, open-label, two-group, two-period crossover study. Cohort 8 will be initiated after Cohorts 1 to 7 are completed.

ELIGIBILITY:
Inclusion Criteria

1. Japanese healthy adult males aged ≥20 and <45 years at the time of informed consent who are non-smokers or able to stop smoking from at least 4 weeks before study drug administration until the post-treatment examination.
2. Has voluntarily consented, in writing, to participate in this study.
3. Has been thoroughly briefed on the conditions for participation in the study, and is willing and able to comply with the conditions.

Exclusion Criteria

1. History of surgical treatment that may affect the pharmacokinetics of the study drug at screening.
2. Suspected to have clinically abnormal symptoms or impairment of organ function requiring treatment on the basis of history and complications at screening, and physical findings, vital signs, ECG findings, or laboratory values at screening or baseline.
3. History of drug allergy at screening.
4. Judged by the investigator or sub-investigator to be inappropriate for participation in this study.

Ages: 20 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2016-09-26 (Actual); Primary Completion 2017-08-17 (Actual); Study Completion 2017-08-17 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment emergent adverse events (TEAEs) and serious adverse events (SAEs) as a measure of safety and tolerability | Days 1 to 14 (Cohort 1 to 7), Days 1 to 21 (Cohort 8)

SECONDARY OUTCOMES:
Maximum observed serum concentration (Cmax) of E6130 | Days 1 to 6 (Cohort 1 to 7), Days 1 to 6 and 8 to 13 (Cohort 8)
Time to Cmax (Tmax) of E6130 | Days 1 to 6 (Cohort 1 to 7), Days 1 to 6 and 8 to 13 (Cohort 8)
Area under the serum concentration-time curve from time zero to time t (AUC(0-t)) of E6130 | Days 1 to 6 (Cohort 1 to 7), Days 1 to 6 and 8 to 13 (Cohort 8)
Area under the serum concentration-time curve from time zero to infinity (AUC(0-inf)) of E6130 | Days 1 to 6 (Cohort 1 to 7), Days 1 to 6 and 8 to 13 (Cohort 8)
Apparent terminal phase half-life (t1/2) of E6130 | Days 1 to 6 (Cohort 1 to 7), Days 1 to 6 and 8 to 13 (Cohort 8)

CONTACTS AND LOCATIONS:
Locations (1):
- Sumida City, Tokyo, Japan